CLINICAL TRIAL: NCT01307085
Title: Effect of Remote Ischemic Preconditioning on Lung Injury in Patients Undergoing Pulmonary Resection:a Randomised Controlled Trial
Brief Title: Effect of Remote Ischemic Preconditioning on Lung Injury After Pulmonary Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cai Li (Other)
Responsible Party: Sponsor-Investigator, Cai Li, Department of Anesthesiology, First Affiliated Hospital, Sun Yat-Sen University, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RIP1126
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Lung Neoplasms
Keywords: remote ischemic preconditioning; lung injury; pulmonary resection
MeSH Terms: conditions — Lung Neoplasms; Lung Injury

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- preconditioning (Experimental): Adult patients undergoing elective pulmonary lobectomy were received a remote ischemic preconditioning group after induction of anaesthesia.
  Interventions: Procedure: remote ischemic preconditioning
- conventional (No Intervention): Adult patients undergoing pulmonary lobectomy were received no treatment after induction of anaesthesia.

INTERVENTIONS:
Procedure: remote ischemic preconditioning — Remote ischaemic preconditioning consisted of three 5-min cycles of right upper limb ischaemia, induced by an automated cuff-inflator placed on the upper arm and inflated to 200 mm Hg, with an intervening 5 min of reperfusion during which the cuff was deflated.
  Other Names: RIP
  Arms: preconditioning

SUMMARY:
The purpose of this study is to determine whether ischemic preconditioning reduces lung injury in patients undergoing pulmonary resection.

DETAILED DESCRIPTION:
Remote ischemic preconditioning is an intervention in which brief ischemia of one tissue or organ protects remote organs from a sustained episode of ischemia. It is known that one-lung ventilation in patients undergoing pulmonary resection, which may cause acute lung injury. The investigators did a single-blinded randomised controlled study to establish whether remote ischemic preconditioning reduces lung injury in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pulmonary carcinoma
* Must be received pulmonary lobectomy

Exclusion Criteria:

* Cardiac disease categorized as NYHA classes II-IV
* Preoperative severe impairment of respiratory function (arterial oxygen tension (PaO2) <60 mmHg or FEV1<50% predicted),
* Pre-existing coagulopathy or thrombocytopenia
* Prior receipt of chemotherapy or radiation therapy or immunotherapy
* Systemic or local active infections (either clinically defined or suggested by evidence such as elevated C-reactive protein levels, leukocytosis, or a body temperature>38℃)
* Peripheral vascular disease affecting the upper limbs
* Administration of vitamins, nonsteroidal anti-inflammatory agent or corticosteroid within 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Limb remote ischemic preconditioning has effective protection of lung injury in patients undergoing pulmonary lobectomy | June,2013
  PaO2/FiO2 in the limb RIPC group was significantly higher than that in the control group at 30 and 60 min after OLV, 30 min and 6 h after operation (all P<0.05)

SECONDARY OUTCOMES:
Cs and Cd | June,2013
  Cs and Cd in limb RIPC group were significantly higher than those in the control group at 30 and 60 min after OLV (all P<0.05)
IL-6 and TNF-α | June,2013
  The IL-6 levels in the limb RIPC group were lower than those in the control group at 30 min, 6, 12, 24 and 48 h after operation (all P<0.05), and there was a significant difference in TNF-α level between the groups (P<0.01).

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Ke Liu, Ph.d, Principal Investigator — Department of Anesthesiology, The First Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Departmeng of Anesthesiology, The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China